CLINICAL TRIAL: NCT05240092
Title: The Effect of Haptonomy Applied to Pregnant Women on Perceived Stress, Fear of Childbirth and Prenatal Attachment
Brief Title: The Effect of Haptonomy Applied to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof. Dr, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SIVAS02
Record Dates: First submitted 2021-12-20; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: First Pregnancy
Keywords: Fear of Childbirth; Haptonomy; Perceived Stress; Prenatal Attachment
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haptonomy Group (Experimental): A home visit was made to the experimental group, and haptonomy was applied for at least 30 minutes, once a week, for 7 weeks (with the researcher for 3 weeks, with the husband by providing the training brochure and video that will help the practice for the next 4 weeks).
  Interventions: Behavioral: Haptonomy
- Standard of care Group (No Intervention): The control group did not receive any treatment.

INTERVENTIONS:
Behavioral: Haptonomy — Haptonomy, as a field dealing with emotional contact through touch, describe the relationship between parents and the unborn baby.
  Other Names: Control Group
  Arms: Haptonomy Group

SUMMARY:
Introduction: Stress experienced during pregnancy can increase fear of childbirth, cause negative perinatal outcomes, and adversely affect the maternal-infant attachment process. This study was conducted to determine the effect of haptonomy applied to pregnant women on perceived stress, fear of childbirth, and prenatal attachment.

Methods: The population of the randomized controlled experimental study consisted of 72 primiparous pregnant women within the gestational weeks 22-28 who presented to the Obstetrics and Gynecology Polyclinic of a state hospital in Turkey for check-up (36 experimental subjects, 36 control subjects).

DETAILED DESCRIPTION:
Background: Stress experienced during pregnancy can increase fear of childbirth, cause negative perinatal outcomes, and adversely affect the maternal-infant attachment process.

Aim: This study was conducted to determine the effect of haptonomy applied to pregnant women on perceived stress, fear of childbirth, and prenatal attachment.

Methods: The population of the randomized controlled experimental study consisted of 72 primiparous pregnant women within the gestational weeks 22-28 who presented to the Obstetrics and Gynecology Polyclinic of a state hospital in Turkey for check-up (36 experimental subjects, 36 control subjects). A home visit was made to the experimental group, and haptonomy was applied for at least 30 minutes, once a week, for 7 weeks (with the researcher for 3 weeks, with the husband by providing the training brochure and video that will help the practice for the next 4 weeks). The control group did not receive any treatment. Data were collected at the first, third, and seventh weeks using the Pregnancy Description form, the Perceived Stress Scale (PSS), the Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A), and the Prenatal Attachment Inventory (PAI). Number and percentage distribution, chi-square test, t test, Mann-Whitney U test, repeated measures, two-way analysis of variance, Friedman test, and Cohen d test were used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women who were married,
* aged 18 years and over,
* literate,
* living in the city center,
* not having any health problems in themselves and their infants,
* with spontaneous pregnancy at 22-28 weeks of gestation,
* without perception and communication problems,
* and who agreed to participate in the study were included in the study.

Exclusion Criteria:

• Multiparity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline
  The PSS is a validated, The scale consists of 10 items, each item receives 1,2,3,4,5 points in turn and is evaluated over total score. Total score ranges from 10-50, and an increase in the score indicates an increase in perceived stress level.
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Baseline
  The W-DEQ-A is a validated,to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Prenatal Attachment Inventory (PAI) | Baseline
  The PSS is a validated, explain thoughts, feelings, and situations experienced by woman during pregnancy and to determine the level of attachment to infant in prenatal period. Each item is of a four-point Likert type, with a score between 1 and 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increase in the score obtained by pregnant indicates that level of attachment also increases.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Week 3
  The PSS is a validated, The scale consists of 10 items, each item receives 1,2,3,4,5 points in turn and is evaluated over total score. Total score ranges from 10-50, and an increase in the score indicates an increase in perceived stress level.
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Week 3
  The W-DEQ-A is a validated,to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Prenatal Attachment Inventory (PAI) | Week 3
  The PSS is a validated, explain thoughts, feelings, and situations experienced by woman during pregnancy and to determine the level of attachment to infant in prenatal period. Each item is of a four-point Likert type, with a score between 1 and 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increase in the score obtained by pregnant indicates that level of attachment also increases.

OTHER OUTCOMES:
Perceived Stress Scale (PSS) | Week 7
  The PSS is a validated, The scale consists of 10 items, each item receives 1,2,3,4,5 points in turn and is evaluated over total score. Total score ranges from 10-50, and an increase in the score indicates an increase in perceived stress level.
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Week 7
  The W-DEQ-A is a validated,to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Prenatal Attachment Inventory (PAI) | Week 7
  The PSS is a validated, explain thoughts, feelings, and situations experienced by woman during pregnancy and to determine the level of attachment to infant in prenatal period. Each item is of a four-point Likert type, with a score between 1 and 4. A minimum score of 21 and a maximum score of 84 can be obtained from the scale. Increase in the score obtained by pregnant indicates that level of attachment also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Sükran Ertekin Pinar, Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Background] Muller ME. Development of the Prenatal Attachment Inventory. West J Nurs Res. 1993 Apr;15(2):199-211; discussion 211-5. doi: 10.1177/019394599301500205. No abstract available. PMID 8470375
- [Background] Veringa IK, de Bruin EI, Bardacke N, Duncan LG, van Steensel FJ, Dirksen CD, Bogels SM. 'I've Changed My Mind', Mindfulness-Based Childbirth and Parenting (MBCP) for pregnant women with a high level of fear of childbirth and their partners: study protocol of the quasi-experimental controlled trial. BMC Psychiatry. 2016 Nov 7;16(1):377. doi: 10.1186/s12888-016-1070-8. PMID 27821151
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- See also: Adam, E. M. (2012). L' haptonomie Un projet pour une naissance. Published online. — https://hal.univ-lorraine.fr/hal-01875566/document
- See also: Arabin, B., & Metz, G. A. S. (2020). Environmental enrichment and pregnancy: paradigms of (epi)genetic effects of social or sensory stimulation. Gynakologe, 53(7), 433-443. https://doi.org/10.1007/s00129-020-04622-2 — https://doi.org/10.1007/s00129-020-04622-2
- See also: Arfaie, K., Nahidi, F., Simbar, M., & Bakhtiari, M. (2017). The role of fear of childbirth in pregnancy related anxiety in Iranian women: a qualitative research. Electronic Physician, 9(2), 3733-3740. https://doi.org/http://dx.doi.org/10.19082/3733 — https://doi.org/http://dx.doi.org/10.19082/3733
- See also: Arslan, A., & Temiz, G. (2019). The knowledge, attitude and behavior levels of midwifery students for the non-pharmacological methods used in the management of labor pain. Perinatal Journal, 27(2), 77-88. https://doi.org/10.2399/prn.19.0272006 — https://doi.org/10.2399/prn.19.0272006
- See also: Célestin-Lhopiteau, I., & Wanquet-Thibault, P. (2018). Haptonomie. In: guide des pratiques psychocorporelles: 25 techniques (relaxation, hypnoseart-thérapie, toucher, etc.) (2nd ed., pp. 186-190). Elsevier Health Sciences. — https://www.elsevier-masson.fr/guide-des-pratiques-psychocorporelles-9782294758584.html
- See also: CIRDH. (2018a). Haptonomie pré et postnatale. International Center for Research and Development of Haptonomy. Published 2018. Accessed November 18, 2020. — https://haptonomie.org/
- See also: CIRDH. (2018b). Presentation of haptonomy: Haptonomy. International center for research and development of haptonomy. Published 2018. Accessed August 28, 2020. — https://www.haptonomie.org/en/
- See also: Dayton, CJ., Brown, S., Goletz, J., Hicks, L., Barron, C., Sperlich, M., & Smith-Darden, J. (2019). Pathways to parenting: predictors of prenatal bonding in a sample of expectant mothers and fathers exposed to contextual risk. — https://doi.org/10.1007/s10826-019-01343-6
- See also: Dencker, A., Nilsson, C., Begley, C., Jangsten, E., Mollberg, M., Patel, H., Wigert, H., Hessman, E., Sjöblom, H., & Sparud-Lundin, C. (2019). Causes and outcomes in studies of fear of childbirth: a systematic review. Women and Birth, 32(2), 99-111. — https://doi.org/10.1016/j.wombi.2018.07.004
- See also: Dereli Yilmaz, S., & Kizilkaya Beji, N. (2013). Prenatal B Turkish version of prenatal attachment inventory: a study of reliability and validity. Journal of Anatolia Nursing and Health Sciensces, 16(2), 103-109. — https://dergipark.org.tr/tr/download/article-file/29648
- See also: Dolto, C. (2018). L'accompagnement pré- et postnatal par l'haptonomie. SoinS Pédiatrie-Puériculture, 39(300), 24-26. — https://doi.org/10.1016/j.spp.2017.11.005
- See also: Erci, B. (2006). Relıabılıty and valıdıty of the turkısh versıon of generalızed perceıved self-effıcacy scale. Ataturk University School of Nursing, 9(1), 58-63. — https://dergipark.org.tr/tr/pub/ataunihem/issue/2632/33865
- See also: Faul, F., Erdfelder, E., Buchner, A., & Lang, A.G. (2009). Statistical power analyses using G*Power 3.1: Tests for correlation and regression analyses. Behavior Research Methods, 41(4), 1149-1160. — https://doi.org/10.3758/BRM.41.4.1149
- See also: Fernández Fernández-Arroyo, M. (2020). Childbirth Education: Comparative Analysis. In M. Z. Jovandaric & S. J. Milenkovic (Eds.), Childbirth (Vol. 32, Issue July, pp. 137-144). IntechOpen. — https://doi.org/10.5772/intechopen.88021
- See also: Hanley, J., Hara, MO., Omay, O., Laure, A., Wisner, K., Coen, A. et. al (2013). The marcé international society international biennial general scientific meeting.Archives of Women's Mental Health, 16(S1), 129 — https://doi.org/10.1007/s00737-013-0355-x
- See also: Hermon, N., Wainstock, T., Sheiner, E., Golan, A., & Walfisch, A. (2019). Impact of maternal depression on perinatal outcomes in hospitalized women-a prospective study. Archives of Women's Mental Health, 22(1), 85-91. — https://doi.org/10.1007/s00737-018-0883-5
- See also: Hobek Akarsu, R., & Rathfisch, G. (2018). The effect of pregnancy yoga on the pregnant's psychosocial health and prenatal attachment. Indian Journal of Traditional Knowledge, 17(4), 732-740. — http://nopr.niscair.res.in/bitstream/123456789/45060/1/IJTK%2017(4)%20732-740.pdf
- See also: Hobek Akarsu, R., Tuncay, B., & Yuzer Alsac, S. (2017). Evidence-based applications in mother-infant attachment. Gumushane University Journal of Health Sciences, 6(4), 275-279. — https://dergipark.org.tr/tr/pub/gumussagbil/issue/32215/370447
- See also: Kaur, M. (2020). Evidence-based applications in mother-infant attachment. Gumushane University Journal of Health Sciences, 8(3), 263-267. — https://doi.org/10.5958/2454-2652.2020.00058.x
- See also: Kemper, H. C. (2017). Haptotherapy and science Revealing the secret of good research designs and valid measurement methods. International Journal of Haptonomy and Haptotherapy, 10(081708), 10-17. — https://ijhh.org/wp-content/uploads/2019/12/2017-08-10-Han-Kemper-Haptotherapy-and-science.pdf
- See also: Klabbers, G. A. (2018). Can haptotherapy reduce fear of childbirth? Some first answers from a randomized controlled trial. Tilburg University. Published online. Netherlands. — https://pure.uvt.nl/ws/portalfiles/portal/27445680/Klabbers_Can_Haptotherapy_05_09_2018_.pdf
- See also: Klabbers, G. A., Paarlberg, K. M., & Vingerhoets, A. J. J. M. (2018). Does haptotherapy benefit mother-child bonding in women with high fear of childbirth? International Journal of Haptonomy and Haptotherapy, 3(1), 1-7. — https://research.tilburguniversity.edu/en/publications/does-haptotherapy-benefit-mother-child-bonding-in-women-with-high
- See also: Klabbers, G. A., van den Heuvel, M. M. A., van Bakel, H. J. A., & Vingerhoets, A. J. J. M. (2016). Severe fear of childbirth: Its features, assesment, prevalence, determinants, consequences and possible treatments. Psychological Topics, 25(1), 107-127. — https://research.tilburguniversity.edu/en/publications/severe-fear-of-childbirth-its-features-assesment-prevalence-deter
- See also: Klabbers, GA., Wijma, K., Paarlberg, KM., Emons, WHM., & Vingerhoets, AJJM. (2014). Treatment of severe fear of childbirth with haptotherapy: Design of a multicenter randomized controlled trial. BMC, 14(1). — https://doi.org/10.1186/1472-6882-14-385
- See also: Koc Ozkan, T., Simsek Kucukkelepce, D., & Aydın Ozkan, S. (2020). Relationship between prenatal attachment and body sense in pregnancy and affecting factors. Manisa Celal Bayar University Journal of Institute of Health Science, 7(1), 49-54. — https://doi.org/10.34087/cbusbed.587467
- See also: Ksycinski, W., Hartman-Ksycinska, A., & Pszeniczna, E. (2010). PP-272. Prenatal baby's behaviour with the use of haptonomic techniques and the relevant experiences and reactions of the parents. Early Human Development, 86, S125. — https://doi.org/10.1016/j.earlhumdev.2010.09.328
- See also: Larsson, B., Karlström, A., Rubertsson, C., Ternström, E., Ekdahl, J., Segebladh, B., & Hildingsson, I. (2017). Birth preference in women undergoing treatment for childbirth fear: A randomised controlled trial. Women and Birth, 30(6), 460-467. — https://doi.org/10.1016/j.wombi.2017.04.004
- See also: Paica, C. I. (2017). Prenatal and postnatal psychological counselling the conscious assumption of the maternal role. Journal of Experiential Psychotherapy, 20(2), 24-31. — https://jep.ro/images/pdf/cuprins_reviste/78_art_4.pdf
- See also: Poirier, P. (2011). La préparation à la naissance et à la parentalité, ce qu'en savent les futurs parents [Université d'Angers]. — https://dune.univ-angers.fr/documents/dune334
- See also: Pollmann, M. T. F., & Hoffenaar, P. J. (2017). Haptonomische zwangerschapsbegeleiding en de prenatale gehechtheid van ouders aan hun kind. Kind En Adolescent, 38(2), 108-119. — https://doi.org/10.1007/s12453-017-0139-6
- See also: Rathfisch, Gulay. (2019). Prenatal haptonomy course notes [PowerPoint slide]. İstanbul. — https://avesis.istanbul.edu.tr/gulay.rathfisch/egitim
- See also: Stojanow, K., Rauchfuss, M., Bergner, A., & Maier, B. (2017). Anxiety in high-and low-risk pregnancies and its influence on perinatal outcome. Mental Health and Prevention, 6, 51-56. — https://doi.org/10.1016/j.mhp.2017.03.001
- See also: Tison, R. B. (2019). L' accompagnement haptonomique prénatal : attentes et vécu des couples. ESF - UCA - École de Sages-Femmes - Clermont-Auvergne. — https://dumas.ccsd.cnrs.fr/dumas-02505621
- See also: Vignoli, L. (2016). Préparation à la naissance et à la parentalité en couple: ce qu'en pensent les primipères. — http://bibnum.univ-lyon1.fr/nuxeo/nxfile/default/e19c6302-d00e-4fc8-a916-2115e3bdb85f/file:content/Msfb_2016_VIGNOLI_Lucie.pdf
- See also: Vinit, F. (2010). Réflexions autour de l'accompagnement haptonomique de la grossesse. Filigrane, 18(2), 38-50. — https://doi.org/10.7202/039288ar
- See also: Woods, S. M., Melville, J. L., Guo, Y., Fan, M., & Gavin, A. (2010). Psychosocial stress during pregnancy. American Journal of Obstetrics & Gynecology, 202(1), 61.e1-61.e7. — https://doi.org/10.1016/j.ajog.2009.07.041